CLINICAL TRIAL: NCT01296880
Title: Effects of Adjunctive Lacosamide on Mood States and Quality of Life (QOL) in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-011
Record Dates: First submitted 2011-02-09; First posted 2011-02-16 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2012-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LCM group: Patients who are having lacosamide (LCM) added to their anti-epileptic drug regimen
- control group: Patients who are NOT having lacosamide (LCM) added to their anti-epileptic drug regimen

SUMMARY:
The purpose of this study is to determine the effect of lacosamide on mood and quality of life in people with epilepsy.

DETAILED DESCRIPTION:
Lacosamide (LCM) was found in phase 3 studies to have good efficacy and tolerability as adjunctive treatment in adult patients with uncontrolled partial onset seizures, with or without secondary generalization. Dose-related adverse drug reactions (ADRs) included dizziness, headache and nausea, but the incidence of reported mood symptoms was similar to placebo. The very low incidence of such events, combined with LCM's unique mechanism of action, suggest that LCM has the potential to be among the few anti-epileptic drugs (AEDs) without clinically significant mood ADRs.

The effects of LCM on mood states (i.e., worsening or improvement) have not been examined with standardized measures. In addition, its effects on quality of life (QOL) have not been explored, although QOL is known to be affected by other AEDs.

The investigators propose to examine the effects of LCM on mood and QOL in a real-world population of adult patients with partial-onset seizures. To the knowledge of the investigators, the proposed study will be the first to examine these domains in a scientifically rigorous fashion in patients treated with LCM. Thus, study results will fill a current knowledge gap, and will provide important information to clinicians and patients when considering LCM treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 17 years old
* Have partial (focal) onset seizures that are not controlled with medication
* (LCM group only) LCM is being added to anti-epileptic drug regimen by treating physician

Exclusion Criteria:

* Have taken LCM in the past.
* Change in anti-epileptic drugs or their doses in the past 28 days.
* Have participated in another drug research study in the past 3 months.
* Have had epilepsy brain surgery, or plan to have epilepsy surgery in the next four months.
* Have a psychiatric or behavioral condition, which in the opinion of the investigator, could compromise patient's ability to participate in the study.
* Have a progressive (worsening) disease that affects patients brain and its functions.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being treated at epilepsy clinics at SUNY Downstate Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in overall Quality of Life in Epilepsy-89 (QOLIE-89) score | baseline and 3 months later
Change from baseline in Profile of Mood States (POMS) score | baseline and 3 months later

SECONDARY OUTCOMES:
Change from baseline in QOLIE-89 subtests | baseline and 3 months later
Change from baseline in POMS subtests | baseline and 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Arthur C Grant, MD, PhD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States